CLINICAL TRIAL: NCT06336941
Title: Intraoral Ultra-High Frequency Ultrasound of Oral Soft Tissue Lesions
Brief Title: "Ultra-High Frequency intraOral UltraSonography of the TONgue" (HOUSTON)
Acronym: HOUSTON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Rossana Izzetti, Researcher at the Department of Surgical, Medical and Molecular Pathology and Critical Care Medicine of the University of Pisa, Principal Investigator, University of Pisa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 32822
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: oral neoplasm; ultrasonography; depth of invasion
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound group (Experimental): The patients with a clinical diagnosis of oral squamous cell carcinoma will undergo intraoral ultrasonographic scan with a 70 MHz frequency probe to evaluate tumor depth of invasion and thickness
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Ultrasonographic scan with a 70 MHz probe

SUMMARY:
Oral diseases are currently diagnosed by means of clinical examination and supported by surgical biopsy procedures. In particular, daily oral medicine practice is lacking the use of a routine diagnostic support to the visualization of anatomical structures located beyond the mucosal surface. Considering the growing interest in minimally invasive diagnosis, the possibility of having an imaging technique dedicated to the investigation of oral soft tissues and their alterations may be instrumental to support the clinical diagnosis. Therefore, attempts to introduce conventional ultrasonography (US) to the diagnostic work-up of pathological conditions of the head and neck have been done, exploiting the unique features of this technique in terms of limited invasive- ness, repeatability, and cost efficiency.

In the literature, both extraoral and intraoral applications of US have been reported. Extraoral applications mainly focus on the characterization of oral and maxillofacial swellings of various origin, while intraoral applications mostly involve the study of malignant lesions in terms of tumor thickness and depth of invasion. The aim of the present protocol is to evaluate the role of intraoral ultra-high frequency ultrasonography in the study of oral mucosal lesions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of oral squamous cell carcinoma
* Eligibility for surgical treatment
* Acceptance to be included in the study

Exclusion Criteria:

* Oral lesions other than oral squamous cell carcinoma
* Pregnant or breastfeeding patients
* Uncontrolled chronic diseases and/or conditions hindering the participation in the study
* Denial of inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-06-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Depth of invasion | measured preoperatively
  Measurement of Depth of invasion on ultrasonography

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Pisa, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No